CLINICAL TRIAL: NCT00675961
Title: Effectiveness of Alcohol Interventions Among TB Patients in Tomsk Oblast, Russia
Brief Title: Effectiveness of Alcohol Interventions Among Tuberculosis (TB) Patients in Tomsk Oblast, Russia
Acronym: IMPACT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Collaborators: Mclean Hospital (Other); Harvard School of Public Health (HSPH) (Other)
Responsible Party: Principal Investigator, Sonya Sunhi Shin, Associate Physician, Brigham and Women's Hospital
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: 2005P-002539; NIH 1 RO1 AA016318-01
Record Dates: First submitted 2008-05-08; First posted 2008-05-12 (Estimated); Last update posted 2017-10-25 (Actual); Status verified 2017-10

CONDITIONS: Tuberculosis; Alcohol Use Disorders
Keywords: Tomsk; TB-Alcohol; Alcohol and co-occurring disease; Brief counseling intervention; Naltrexone
MeSH Terms: conditions — Tuberculosis; Alcoholism | interventions — Naltrexone; 2-benzylidene-3-(cyclohexylamino)-2,3-dihydro-1H-inden-1-one; Therapeutics

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- 1 (Experimental): Behavioral Counseling Intervention (BCI) plus treatment as usual (TAU) (i.e. standard referral to and management by an addictions specialist)
  Interventions: Behavioral: Brief Counseling Intervention (BCI)
- 2 (Experimental): Naltrexone/ Brief Behavioral Compliance Enhancement Treatment (BBCET) plus TAU
  Interventions: Drug: Naltrexone
- 3 (Experimental): BCI + Naltrexone/BBCET plus TAU
  Interventions: Other: BCI + Naltrexone
- 4 (Active Comparator): Treatment as Usual (TAU)
  Interventions: Behavioral: Treatment as Usual

INTERVENTIONS:
Behavioral: Brief Counseling Intervention (BCI) — Two-tiered BCI characterized by both primary and secondary interventions. Primary BCI treatment format consists of 6 discussions delivered monthly in the first 6 months of standard TB treatment. 10-15 minutes long. Secondary BCI is delivered on a monthly basis while receiving TB treatment. 5-10 minutes long.
  Arms: 1
Drug: Naltrexone — Opioid antagonist, which decreases the pleasurable response to and craving for alcohol consumption. Oral; single daily dose of 50 mg per day for 6 months.
  Arms: 2
Other: BCI + Naltrexone — Combination of the two previous interventions
  Arms: 3
Behavioral: Treatment as Usual — Services provided by psychologists and narcologists (additions specialists) employed by the Tomsk Oblast TB Services.
  Arms: 4

SUMMARY:
The primary goal of this study is to assess the effectiveness of two alcohol interventions administered singly or in combination as an integrated component of TB care provided to patients with co-occurring TB and AUDs in Tomsk, Russia. Here we propose two parts of this study:

First, a pilot study to provide Naltrexone to TB patients will be conducted. If feasibility and safety are demonstrated, then we will conduct a randomized clinical trial (RCT) of the following four study arms:

1. A Behavioral Counseling Intervention (BCI) plus treatment as usual (TAU) (i.e. standard referral to and management by an addictions specialist);
2. Naltrexone/ Brief Behavioral Compliance Enhancement Treatment (BBCET) plus TAU
3. BCI + Naltrexone/BBCET plus TAU
4. TAU The RCT will be conducted only if Naltrexone use proves safe and feasible in the pilot study. However, because the pilot does not have a control group and nor is it a Phase I clinical trial, we define "safety" here as demonstration of appropriate adverse event management and adequate safety monitoring procedures, all of which will also be used in the RCT.

The specific aims of the pilot are:

1. To determine the feasibility of administering Naltrexone to patients receiving TB treatment, and
2. To assess the safety of administering Naltrexone to patients receiving TB treatment.

The investigators aim to test the following hypotheses for the pilot: co-administration of Naltrexone with TB treatment is feasible and safe in a population of TB patients with AUDs.

The specific aims of the RCT are:

1. To compare TB treatment outcomes among patients in each of the three intervention arms with the control arm of treatment as usual, and
2. To compare the change in mean number of heavy drinking days in last month of study period compared with baseline among patients in each of the three intervention arms with the control arm of treatment as usual.

The investigators aim to test the following hypotheses for the RCT: Individuals receiving one of the three interventions (Naltrexone, BCI or the combination of Naltrexone/BCI) will experience better TB outcomes and a greater change in the mean number of heavy drinking days, compared with individuals receiving treatment as usual.

DETAILED DESCRIPTION:
An important aspect of the delivery of these alcohol interventions will be their incorporation into TB care and delivery by non-alcohol specialists, i.e. TB physicians. In this study, we propose to exploit the strengths of the TB care delivery paradigm (DOTS) by linking to this care system the provision of alcohol interventions. In order to develop this integrated system, we propose the following innovative approaches to AUD management among TB patients:

1. The Behavioral Counseling Intervention (BCI) will be adapted through iterative collaboration of an interdisciplinary team of local and international specialists to derive a protocol that is easily integrated into routine patient care by TB physicians. This process will include assessment for feasibility and cultural acceptability within the Tomsk clinic and the evaluation of TB physicians for adherence to the BCI protocol.
2. Secondary interventions, incentives and case management, will be implemented to maximize the primary BCI intervention delivered by the TB physician and increase patient motivation to change drinking behavior. These will be designed to capitalize on similar case holding strategies already in place in the Tomsk TB services.
3. Naltrexone will be delivered in the context of DOTS, administered under direct observation administration along with TB medications.

To our knowledge, this is the first study to examine the feasibility of alcohol care when delivered as part of routine TB care and to assess this treatment model's impact on both TB and alcohol outcomes. If proven feasible and effective, this treatment model could be adapted for patients with AUDs and co-occurring medical conditions in other settings. First, this model could be used anywhere co-occurring AUDs adversely affect TB outcomes, including the United States. Second, this strategy could integrate alcohol treatment with medical care of other chronic conditions that are affected by poor adherence due to alcohol use. In particular, the greatest global challenge to treating HIV infection in populations with high rates of substance use is the successful management of substance use to ensure adherence to antiretroviral therapy.

ELIGIBILITY:
Inclusion Criteria:

* Are newly diagnosed with Pulmonary TB: infiltrative, disseminated, or other forms of TB in phase of disintegration
* Will initiate TB treatment in one of 7 study sites (Tomsk Oblast TB Hospital, polyclinic, day hospital, and raions)
* Are 18 years and older
* Are diagnosed with alcohol abuse and dependence by the CIDI-SAM; and
* Signed informed consent

Exclusion Criteria:

* Have liver function tests more than 3x the upper limit of normal range. The participant can be retested after 5 days; if any of the repeat liver function tests is more than 3x upper limit of normal range, the person is excluded
* Reported opioid use in the past month or positive during screen for opioids. The participant can be retested after 5 days; if the second urine screen is positive, the person is excluded;
* Are pregnant or breastfeeding;
* Demonstrate inadequate understanding of the study after undergoing informed consent; or
* Have any co-occurring other medical or psychiatric condition that would make it impossible for them to comply with the study procedures.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Actual)
Dates: Start 2007-01; Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
Alcohol: change in mean number of heavy drinking days in last month of study period compared with baseline | 6 months
TB: successful treatment vs. non-successful treatment as defined by the WHO | 6 months

SECONDARY OUTCOMES:
Time to death | 6 months
Nonadherence to TB therapy, defined as having taken less than 80% of indicated doses | 6 months
Acquisition of drug resistance, defined as new resistance confirmed by DST performed during the study period (compared with baseline DST) to any TB drug to which the subject was exposed during the study | 6 months
Change in the mean number of heavy drinking days (defined as 4 drinks per drinking day for women and 5 drinks per drinking day for men) in the last month of the study compared with baseline | 6 months
Change in mean Addiction Severity Index (ASI) alcohol scores at the end of the study period, compared with baseline | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Sonya S Shin, MD, MPH, Principal Investigator — Division of Global Health Equity, Brigham and Women's Hospital; Harvard Medical School; Viktoriya Livchits, MD, MSc, Study Director — Division of Global Health Equity, Brigham and Women's Hospital; Partners In Health
Locations (1):
- Tomsk Oblast TB Services, Tomsk, Tomsk Oblast, Russia

REFERENCES:
- [Derived] Greene MC, Kane J, Alto M, Giusto A, Lovero K, Stockton M, McClendon J, Nicholson T, Wainberg ML, Johnson RM, Tol WA. Psychosocial and pharmacologic interventions to reduce harmful alcohol use in low- and middle-income countries. Cochrane Database Syst Rev. 2023 May 9;5(5):CD013350. doi: 10.1002/14651858.CD013350.pub2. PMID 37158538
- [Derived] Miller AC, Nelson AK, Livchits V, Greenfield SF, Yanova G, Yanov S, Connery HS, Atwood S, Lastimoso CS, Shin SS; Tomsk Tuberculosis Alcohol Working Group. Understanding HIV Risk Behavior among Tuberculosis Patients with Alcohol Use Disorders in Tomsk, Russian Federation. PLoS One. 2016 Feb 12;11(2):e0148910. doi: 10.1371/journal.pone.0148910. eCollection 2016. PMID 26871943
- [Derived] Connery H, Greenfield S, Livchits V, McGrady L, Patrick N, Lastimoso CS, Heney JH, Nelson AK, Shields A, Stepanova YP, Petrova LY, Anastasov OV, Novoseltseva OI, Shin SS. Training and fidelity monitoring of alcohol treatment interventions integrated into routine tuberculosis care in Tomsk, Russia: the IMPACT Effectiveness Trial. Subst Use Misuse. 2013 Jun;48(9):784-92. doi: 10.3109/10826084.2013.793715. Epub 2013 Jun 10. PMID 23750742